CLINICAL TRIAL: NCT03317769
Title: Creating Live Interactions to Mitigate Barriers (CLIMB): A Mobile Intervention to Improve Social Functioning in People With Schizophrenia
Brief Title: Creating Live Interactions to Mitigate Barriers
Acronym: CLIMB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSC-1013-17
Record Dates: First submitted 2017-10-18; First posted 2017-10-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Treatment (Experimental): Computerized cognitive training for 18 hours and structured social skills training for 9 hours over a 9 week period.
  Interventions: Other: Computerized Plasticity-Based Adaptive Cognitive Training; Other: Optimized social skills training
- Active Comparator (Active Comparator): Commercially-available computerized training for 18 hours and 9 hours of unstructured support group sessions over a 9 week period.
  Interventions: Other: Commercially available computerized training; Other: Unstructured support group sessions

INTERVENTIONS:
Other: Computerized Plasticity-Based Adaptive Cognitive Training — Training on computerized exercises that targets social cognition for 2 hours per week.
  Arms: Experimental Treatment
Other: Commercially available computerized training — Training on computerized, casual video games for 2 hours per week.
  Arms: Active Comparator
Other: Optimized social skills training — Group-video calls with Specialist for 1 hour per week where participants can interact with Specialist individually or as a group. Specialist will provide guidance, support and feedback, and send links and articles about information and topics discussed during the video calls.
  Arms: Experimental Treatment
Other: Unstructured support group sessions — Unstructured support group-video calls for 1 hour per week. The Specialist will not engage with participants (eg. providing participants with links to articles and additional support) or provide guidance for the group discussion.
  Arms: Active Comparator

SUMMARY:
This study is a validation study to evaluate the acceptability, feasibility and impact of a mobile psychosocial intervention to enhance social functioning in people with schizophrenia.

DETAILED DESCRIPTION:
The goal of this study is to employ an innovative and evidence-based mobile intervention that includes a neuroscience-informed computerized social cognition training program, a Health Insurance Portability and Accountability Act-compliant videoconferencing tool that we will use for psychoeducational group therapy, and peer-to-peer secure social networking for individuals with schizophrenia, in a parallel arm, double-blind, randomized, controlled clinical trial to assess feasibility and initial efficacy, to investigate the intervention's effects on symptoms, social cognition, and quality of life, and to prepare for a large-scale efficacy trial in adults with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a clinical diagnosis of Schizophrenia as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) and confirmed by the Structured Clinical Interview for DSM-5 (SCID)
* Participant must be clinically stable (outpatient status for at least 2 months) at time of screening
* Participants taking psychiatric medications must be on a stable medication regimen for greater than or equal to 4 weeks prior to screening
* Participant must be a fluent English speaker
* Participant must have adequate sensorimotor capacity to perform the program, including visual capacity adequate to read from a computer screen at a normal viewing distance, auditory capacity adequate to understand normal speech, and motor capacity adequate to control a computer mouse
* Participants must be able to use iOS mobile applications

Exclusion Criteria:

* Participants with unstable and/or untreated conditions that may affect cognition, including substance abuse/dependence disorders, cardiovascular, endocrine, neurologic disorder, epilepsy, recent hospitalization, ongoing chemotherapy or other cancer treatment
* Participant has a history of mental retardation, pervasive developmental disorder, head trauma, traumatic brain injury, or other neurological disorder that impairs cognition
* Participants who have had psychiatric hospitalizations in the 8 weeks prior to randomization
* Participants had significant medication or clinical status changes, or adjustment in their antipsychotic treatment in the 4 weeks prior to randomization
* Participants with active suicidal ideations and/or behaviors as measured by the Columbia-Suicide Severity Rating Scale (C-SSRS)
* Participants showing signs of intoxication due to current substance abuse (including alcohol and/or illegal drugs) during any in person visit
* Participants with problems performing assessments or comprehending or following spoken instructions
* Participants enrolled in a concurrent clinical trial involving an investigational pharmaceutical, nutraceutical, medical device, or behavioral treatment that could affect the outcome of this study
* Participant is using computer-based cognitive training programs or has used it within a month of the consent date

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Social Functioning utilizing the Social Functioning Scale. | At 9 weeks
  Between-group magnitude of change in social functioning utilizing the Social Functioning Scale. The Social Functioning Scale (SFS) was constructed specifically to tap areas of social functioning that are crucial to the community maintenance of individuals with schizophrenia. The 7 domains include: social engagement/withdrawal, interpersonal behavior, pro-social activities, recreation, independence-competence, independence-performance, and employment/occupation. The raw scores for each domain are converted to scaled scores, with a mean of 100 and a standard deviation of 15. Higher scores are indicative of greater social functioning.
Negative Symptoms utilizing the Positive and Negative Syndrome Scale. | At 9 weeks
  Between-group magnitude of change in negative symptoms utilizing the Positive and Negative Syndrome Scale. The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of patients with schizophrenia. A rating from 1 to 7 is given to each of the 30 different symptoms. The 7-point rating represents increasing levels of psychopathology: 1= absent, 2=minimal, 3=mild, 4=moderate, 5=moderate severe, 6=severe, and 7=extreme. Of the 30 items included in the PANSS, 7 constitute a Positive Scale, 7 a Negative Scale, and the remaining 16 a General Psychopathology Scale. The scores for these scales are arrived at by summation of ratings across component items. Therefore, the potential ranges are 7 to 49 for the Positive and Negative Scales, and 16 to 112 for the General Psychopathology Scale. Higher scores are indicative of greater symptomatology.
Quality of Life utilizing the Abbreviated Quality of Life Scale. | At 9 weeks
  Between-group magnitude of change in quality of life utilizing the Abbreviated Quality of Life Scale. The Quality of Life Scale (QLS) is a scale commonly used as a measure of functioning in schizophrenia. The Abbreviated QLS (aQLS) includes 7 items representing all four interdependent theoretical constructs of the original 21-item QLS. Behavioral anchors are presented for each item, scored on a 0 (severe impairment) to 6 (high functioning) scale. Higher scores are indicative of greater quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Biagianti, MD, PhD, Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States